CLINICAL TRIAL: NCT00531180
Title: Phase II Trial Comparing 4-Dimensional Computed Tomography Derived Ventilation Versus SPECT/CT Tc-99m Aerosol Ventilation in Patients With Thoracic Malignancies
Brief Title: 4-Dimensional CT Derived Ventilation Versus SPECT Aerosol Ventilation in Patients With Thoracic Malignancies
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2006-0698; R21CA128230 (NIH)
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Esophageal Cancer; Lung Cancer
Keywords: Esophageal Cancer; Lung Cancer; Thoracic Malignancies; 4D CT scans; Lung Function
MeSH Terms: conditions — Esophageal Neoplasms; Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 4-DCT Ventilation Validation (Experimental)
  Interventions: Procedure: 4D CT scans; Procedure: Lung Function Imaging

INTERVENTIONS:
Procedure: 4D CT scans — Three 4D CT scans will be performed. After you are out of the CT scanner, ventilation images will be calculated from the 4D CT images and will be compared with the standard ventilation imaging method.
Procedure: Lung Function Imaging — Lung function imaging performed to provide information on how well the lungs work, how air moves into the lungs with breathing, and blood circulation into the lungs.

SUMMARY:
Objectives:

Primary Objective:

1. To determine the correlation between 4-dimensional computed tomography (4D CT) derived ventilation and single photon emission tomography (SPECT) aerosol Tc-99m determined ventilation.

Secondary Objective:

1. To evaluate the reproducibility of the 4D CT derived ventilation and to obtain an estimate of the variance in a single setting.
2. To assess the correlation between hypoperfused and hypoventilated pulmonary regions in patients with thoracic malignancies.
3. To investigate the effect of continuous positive airway pressure (CPAP) on ventilation and tumor motion.

DETAILED DESCRIPTION:
By using a 4-dimensional (4D) computed tomography (CT) scans researchers will create ventilation (circulation of air) calculations. This new calculation method is quicker and may produce better images than the standard ventilation calculations.

If you agree to take part in this study and are found to be eligible, you will have lung function imaging. Lung function imaging gives researchers information on how well the lungs work, how air moves into the lungs with breathing, and blood circulation into the lungs.

You will have three 4D CT scans performed while you are breathing quietly. A 2-inch plastic box will be placed on top of your chest to monitor the motion of your chest during the scanning. After you are out of the CT scanner (once the scanning is finished), ventilation images are calculated from the 4D CT images and will be compared with the standard ventilation imaging method. The 4D CT imaging will take about 30 minutes to complete.

As part of standard care, once you have finished the 4D CT scan, you will have a single photon emission computed tomography (SPECT) pulmonary (lung) ventilation scan performed. The SPECT ventilation scan requires that you first breathe in a radioactive aerosol (or mist, called Tc-99m DPTA), which will help the study doctor tell where air goes when you breathe. Then you will be placed in the SPECT scanner, and images will be taken of your lungs. The SPECT imaging will take about 1 hour to complete.

Within 10 days after the first imaging session, you will return for a second imaging session. During the second imaging session, you will have a standard of care SPECT pulmonary perfusion (blood supply to tissue and organs) test done. During this test, a radioactive substance is given by vein (called Tc-99m MAA). This substance will get trapped in the lungs, and the SPECT imaging will show the blood flow in the lungs. This test should take 45-60 minutes to complete.

Once you complete the second imaging session, your participation will over in this study.

This is an investigational study. All of the imaging scans used in this study are FDA approved and commercially available. The calculation of ventilation images from 4D CT scanning is investigational and authorized for use in research only. Up to 36 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with pathologic diagnosis of esophagus or lung cancer (Stage I through IV).
2. Patients must be able to lie flat for the duration of the treatment planning sessions.
3. Patients must sign informed consent.
4. Patients who are scheduled to receive radiation therapy.
5. A cohort of 6 lung cancer patients whose primary tumors move greater than 1 cm will be recruited (CPAP cohort).

Exclusion Criteria:

1. Significant pleural effusion as evaluated by the attending Radiation Oncologist is excluded.
2. Women of childbearing potential (A woman of child-bearing potential is a sexually mature woman who has not undergone a hysterectomy or who has not been naturally postmenopausal for at least 24 consecutive months [i.e., who has had menses at any time in the preceding 24 consecutive months]) and male participants must practice effective contraception (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study.
3. Patients with severe COPD or asthma will be excluded from the CPAP cohort.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2007-08-21 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Correlation between 4-dimensional computed tomography (4D CT) derived ventilation and single photon emission tomography (SPECT) aerosol Tc-99m determined ventilation | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heath Skinner, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org